CLINICAL TRIAL: NCT03067610
Title: A Prospective Phase II Study of Involved Field Elective Volume De-Intensification for Oropharyngeal and Laryngeal Squamous Cell Carcinoma Treated With Intensity Modulated Radiation Therapy
Brief Title: Involved Field Elective Volume De-Intensification Radiation Therapy for Head and Neck Cancer
Acronym: INFIELD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David Sher, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 052016-044
Record Dates: First submitted 2016-11-18; First posted 2017-03-01 (Actual); Results first posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Cancer; Carcinoma, Squamous Cell; Neoplasms, Oral; Neoplasms, Pharyngeal
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Mouth Neoplasms; Pharyngeal Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Drug Therapy; Cisplatin; Cetuximab

STUDY DESIGN:
Intervention Model Description: radiation therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiation Therapy (Experimental): Intensity modulated radiation therapy (IMRT) with or without chemotherapy (if given, either cisplatin, cetuximab, or carboplatin-paclitaxel)
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Drug: chemotherapy

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy — The radiotherapy plan wil be delivered in 2 sequential courses. The first course involves 20 fractions of 2 Gy per fraction to the entire volume (gross disease and elective). The second course involves 15 fractions (thus, total of 35 fractions), at either 2 Gy (gross disease) or 1.6 Gy (microscopic disease and suspicious node) per fraction.
  Other Names: IMRT
Drug: chemotherapy — chemotherapy (if given, either cisplatin, cetuximab, or carboplatin-paclitaxel) per physician discretion
  Other Names: cisplatin, cetuximab, or carboplatin-paclitaxel

SUMMARY:
Intensity modulated radiation therapy (IMRT) with or without chemotherapy (if given, either cisplatin, cetuximab, or carboplatin-paclitaxel)

DETAILED DESCRIPTION:
This study aims to significantly improve the acute and late morbidity of patients with oropharyngeal and laryngeal squamous cell carcinoma both by tailoring the elective irradiation only to regions with a legitimate risk of recurrence (> 5%) and by lowering the elective dose to 40 Gy. Level IB will not be electively treated unless it is involved with pathologic or suspicious lymphadenopathy. Level V will not be treated unless two or more ipsilateral nodal levels are involved (or level V itself has pathologic or suspicious adenopathy). Levels III and IV will only be irradiated if the immediately proximal level contains pathologic lymphadenopathy (i.e. level III irradiated if level II is positive; level IV irradiated if level III is positive). We anticipate that this approach should dramatically improve the acute and late complication profile.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-proven diagnosis of squamous cell carcinoma of the oropharynx or larynx. Squamous cell carcinoma of unknown primary is not allowed.
* Patients must have clinically or radiographically evident measureable disease at the primary site and/or nodal stations. Patients may undergo a diagnostic tonsillectomy, and diagnostic lymph node excision (< 2 nodes) is also allowable.
* Clinical stage I-IVB (AJCC, 7th edition); stages I-II glottic cancer are excluded
* Age ≥ 18 years.
* ECOG Performance Status 0-2
* Adequate organ and marrow function as defined below:
* leukocytes ≥ 3,000/mcL
* absolute neutrophil count ≥ 1,500/mcL
* platelets ≥ 100,000/mcl
* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SPGT) ≤ 2.5 X institutional upper limit of normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Negative serum or urine pregnancy test within 2 weeks before registration for women of childbearing potential.
* Neck CT and/or neck MRI, and whole body PET-CT.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Distant metastasis or adenopathy below the clavicles.
* Inability to undergo PET-CT.
* Stage I and II glottic carcinoma.
* Gross total excision of both the primary and nodal disease.
* Synchronous primaries outside of the oropharynx and larynx.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease-free for a minimum of 1 years
* Prior systemic chemotherapy for the study cancer; prior chemotherapy for a remote cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation fields.
* Subjects may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the chemotherapy agents in this study (if necessary).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* History of immunosuppression or autoimmunity, including HIV, and organ or stem cell transplant, or an autoimmune condition previously treated with immunosuppressive therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sher, MD, MPH, Principal Investigator — U Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - University of Texas Southwestern Medical Center - Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy: Intensity modulated radiation therapy (IMRT) with or without chemotherapy (if given, either cisplatin, cetuximab, or carboplatin-paclitaxel). There was only one study arm. The radiation field and dose are the same with or without chemotherapy. The intent is to assess the effects of radiation therapy, regardless of chemotherapy treatment.
  Intensity Modulated Radiation Therapy: The radiotherapy plan wil be delivered in 2 sequential courses. The first course involves 20 fractions of 2 Gy per fraction to the entire volume (gross disease and elective). The second course involves 15 fractions (thus, total of 35 fractions), at either 2 Gy (gross disease) or 1.6 Gy (microscopic disease and suspicious node) per fraction.
  chemotherapy: chemotherapy (if given, either cisplatin, cetuximab, or carboplatin-paclitaxel) per physician discretion
Period: Overall Study
Arm/Group | Radiation Therapy
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 58
  Black | 8
  Hispanic | 4
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 72
Disease site [Count of Participants; unit: Participants]
  Oropharynx | 51
  Larynx | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Solitary Elective Volume Recurrence
Description: The crude risk of 2-year solitary elective volume recurrence will be calculated among all patients who are followed for at least 2 years. Patients who die before 2 years without an SEVR will be included in the denominator.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 72
Participants | 0

2. Secondary Outcome: Quality of Life (QOL) Patient Reported Outcomes (PRO)
Description: Quality of life (QOL) patient-reported outcomes (PRO) for overall number of participants following treatment with elective volume and dose de-escalation, using European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30), EORTC HN35, which is specific to head and neck cancer, and composite MD Anderson Dysphagia Inventory (MDADI).
  EORTC QLQ-C30 and QLQ-H&N35 are scored on a 4-point categorical scale ranging from 1 "not at all" to 4 "very much". This scale is then linearly transformed to a 0-100 scale, where a higher score represents a higher response level. A high score for a functional scale represents higher level functioning, a high score for quality of life represents a high quality of life, and a high score for a symptom scale represents worse symptoms.
  MD Anderson Dysphagia Inventory (MDADI) questionnaire: Possible score ranges from 0-100, with higher score indicating higher functioning.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Total Cohort Baseline: Intensity modulated radiation therapy (IMRT) with or without chemotherapy (if given, either cisplatin, cetuximab, or carboplatin-paclitaxel)
  Intensity Modulated Radiation Therapy: The radiotherapy plan wil be delivered in 2 sequential courses. The first course involves 20 fractions of 2 Gy per fraction to the entire volume (gross disease and elective). The second course involves 15 fractions (thus, total of 35 fractions), at either 2 Gy (gross disease) or 1.6 Gy (microscopic disease and suspicious node) per fraction.
  chemotherapy: chemotherapy (if given, either cisplatin, cetuximab, or carboplatin-paclitaxel) per physician discretion
- Total Cohort 3 Month; Total Cohort 6 Month; Total Cohort 12 Month: Total cohort
Arm/Group | Total Cohort Baseline | Total Cohort 3 Month | Total Cohort 6 Month | Total Cohort 12 Month
Number analyzed (Participants) | 72 | 57 | 44 | 43
score on a scale
  EORTC QLQ30 global | 71.4 (2.3) | 76.9 (2.6) | 79.2 (2.8) | 85.9 (2.3)
  EORTC QLQ30 physical fcn | 90.3 (1.7) | 87.4 (2.3) | 90.3 (2.4) | 93.0 (1.8)
  EORTC QLQ30 role fcn | 81.9 (3.0) | 82.5 (3.4) | 85.6 (3.6) | 95.3 (2.2)
  EORTC QLQ30 emotional fcn | 78.0 (2.8) | 87.7 (2.7) | 82.9 (3.7) | 88.2 (3.2)
  EORTC QLQ30 cognitive fcn | 90.0 (1.9) | 89.5 (2.7) | 86.4 (3.1) | 90.7 (2.9)
  EORTC QLQ30 social fcn | 85.2 (2.4) | 85.1 (3.5) | 85.6 (3.7) | 90.3 (3.4)
  EORTC HN35 dry mouth | 14.4 (2.8) | 59.0 (4.1) | 47.7 (4.5) | 38.0 (4.2)
  EORTC HN35 sticky saliva | 15.7 (3.2) | 38.0 (4.4) | 27.3 (4.4) | 27.1 (4.6)
  EORTC HN35 senses | 6.7 (1.8) | 25.7 (2.9) | 20.1 (3.3) | 15.9 (2.7)
  EORTC HN35 pain | 24.4 (2.7) | 16.5 (2.7) | 14.2 (3.3) | 7.9 (2.3)
  EORTC HN35 speech | 18.4 (2.9) | 13.4 (2.6) | 19.2 (4.5) | 9.8 (2.6)
  Composite MDADI | 81.3 (1.9) | 79.6 (2.0) | 76.9 (2.6) | 84.9 (2.3)

3. Secondary Outcome: Number of Participants With Definite, Possible, and Probable Protocol-related Toxicities (Grade 3-5)
Description: Only adverse events (grade 3-5) assessed to be definitely, probably, or possibly related to protocol treatment up to 2 years post-treatment will be considered. This was measured according to NCI's CTCAE v4.0 toxicity criteria.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 33
Participants | 3

4. Secondary Outcome: Total Number of Participants With Gastrostomy Dependence
Description: The prevalence of gastrostomy use up to 2 years will be described.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 72
Participants | 31

5. Secondary Outcome: Patient Utilities
Description: The average patient utilities (derived from EQ-5D) from baseline up to 2 years from the end of treatment will be described. Changes in patient utility will be analyzed using generalized estimated equations (GEE).
Time Frame: 2 years
Population: Collected data were not considered valid due to software limitations as it was not available to auto-calculate the data as proposed by our EMR
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Description: Overall survival will be calculated from the initiation of treatment using the Kaplan-Meier method.
Time Frame: 2 years
Population: Reported the percentage of the total patient population who survived to 2 years post-treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 72
percentage of patients | 89

7. Secondary Outcome: Progression-free Survival
Description: Progression-free survival will be calculated from the initiation of treatment. Progression is confirmed by biopsy, which will be used as the date of progression.
Time Frame: 2 year
Population: Percentage of the total patient population with progression-free survival 2 years post treatment
Measure: Number; unit: percentage of patients
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 72
percentage of patients | 79

8. Secondary Outcome: Probability of Locoregional or Distant Tumor Failure
Description: The percentage of patients with locoregional or distant failure within 2 years of treatment will be estimated using cumulative incidence statistics, with death serving as the competing risk. Cumulative incidence refers to the estimated risk/probability of tumor failure within 2 years of treatment, either locoregional recurrence or distant metastasis, accounting for the competing risk of death.
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Radiation Therapy
Number analyzed (Participants) | 72
percentage of patients
  Locoregional recurrence | 14
  Distant metastasis | 14

ADVERSE EVENTS:
Time Frame: 30 months
Arm/Group | Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 1/72
Serious Adverse Events (participants affected / at risk) | 35/72
Other Adverse Events (participants affected / at risk) | 65/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (N=72)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Acute Encephalopathy (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (3)
acute mescenteric ischemia (Vascular disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (7)
aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atypical Chest Pain (General disorders) | 1 (1)
chills (General disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 8 (8)
Delirium (Psychiatric disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (1)
dizziness (Nervous system disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 14 (14)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
fatigue (General disorders) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
fever (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypercapnic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 2 (2)
hypotensive (Vascular disorders) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
nausea (Gastrointestinal disorders) | 4 (4)
Neoplasm of unknown etiology (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neutropenic Fever (General disorders) | 1 (1)
Opioid Overdose (General disorders) | 1 (1)
Oral Hemorrhage (Gastrointestinal disorders) | 2 (2)
Oral Mucositis (Gastrointestinal disorders) | 2 (2)
parethesia (Nervous system disorders) | 1 (1)
Radiation Dermatitis (Injury, poisoning and procedural complications) | 1 (1)
seizure (Nervous system disorders) | 1 (1)
sepsis (Infections and infestations) | 2 (2)
Severe systemic inflammatory response syndrome (General disorders) | 1 (1)
Skin infection (cellulitis ) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (N=72)
Abdominal distension (Gastrointestinal disorders) | 1
abdominal pain (Gastrointestinal disorders) | 18
abscess of chin (General disorders) | 1
Acid Reflex (Gastrointestinal disorders) | 11
acne vulgaris (Skin and subcutaneous tissue disorders) | 1 (1)
Acneform rash (Skin and subcutaneous tissue disorders) | 1 (1)
agitated (Psychiatric disorders) | 1 (1)
Albumin Decreased (Metabolism and nutrition disorders) | 1 (1)
alkaline phosphate decreased (Investigations) | 3 (3)
alkaline phosphatase increased (Investigations) | 2 (2)
Allergic Reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 (6)
alopecia (Skin and subcutaneous tissue disorders) | 1
ALP increased (Investigations) | 2
ALT decreased (Investigations) | 3
ALT increased (Investigations) | 11
altered mental status (General disorders) | 4
altered sensation (Nervous system disorders) | 2
Anaerobic infection (Infections and infestations) | 1
anemia (Blood and lymphatic system disorders) | 45 (115)
Anorexia (Metabolism and nutrition disorders) | 25 (30)
anxiety (Psychiatric disorders) | 20 (23)
Aortic injury (Injury, poisoning and procedural complications) | 1
aphonia (Nervous system disorders) | 1
appetite change (Gastrointestinal disorders) | 2
Arm pain (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
aspiration (Respiratory, thoracic and mediastinal disorders) | 7 (8)
AST increased (Investigations) | 7 (9)
asthenia (General disorders) | 1
asthma (Respiratory, thoracic and mediastinal disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Atypical Chest Pain (General disorders) | 2
AV block 1st Degree (Vascular disorders) | 1
Azotemia (Investigations) | 1
back pain (Musculoskeletal and connective tissue disorders) | 15
BCC Nose (General disorders) | 1
bite wound (General disorders) | 1
bladder incontinence (Renal and urinary disorders) | 1
bleeding from mouth (General disorders) | 1
blurred vision (Eye disorders) | 10 (11)
Bloating (Gastrointestinal disorders) | 3
bloody secretion (Vascular disorders) | 2
blurred vision (Eye disorders) | 11
bowel incontinence (Gastrointestinal disorders) | 1
Bradycardia (Cardiac disorders) | 1
breast pain (Hepatobiliary disorders) | 1
breast swelling (General disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Coronary Artery Disease (Cardiac disorders) | 2
calcium count increased (Investigations) | 1
Cardiac troponin I increased (Investigations) | 1
Cellulitis (Infections and infestations) | 2
cervical stenosis of spine (Musculoskeletal and connective tissue disorders) | 1
cervicalgia (Musculoskeletal and connective tissue disorders) | 1
change in mole (Skin and subcutaneous tissue disorders) | 2
Cheilitis (Gastrointestinal disorders) | 1
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1
chest pain (General disorders) | 6
chest tightness (General disorders) | 1
chest wall pain (Cardiac disorders) | 1
chills (General disorders) | 5
Chronic Kidney Disease (Renal and urinary disorders) | 3
Cold Intolerance (General disorders) | 8
confusion (Psychiatric disorders) | 4
congestion (Respiratory, thoracic and mediastinal disorders) | 4
constipation (Gastrointestinal disorders) | 55
contact dermatitis (Skin and subcutaneous tissue disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 24
creatinine decreased (Investigations) | 7
creatinine increased (Investigations) | 15
cystitis (Renal and urinary disorders) | 1
decreased appetite (Metabolism and nutrition disorders) | 3
Decreased platelet count (Investigations) | 2
decreased urine output (Renal and urinary disorders) | 1
decreased WBC (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 27
dental infection (Infections and infestations) | 1
depression (Psychiatric disorders) | 15
dermatitis (Skin and subcutaneous tissue disorders) | 1
Diabetes (Metabolism and nutrition disorders) | 3
diaphoresis (Metabolism and nutrition disorders) | 9
Diarrhea (Gastrointestinal disorders) | 24
discoloration of tongue (Skin and subcutaneous tissue disorders) | 1
Discolored discharge (General disorders) | 1
dizziness (Nervous system disorders) | 21
double vision (Eye disorders) | 1
dry cough (Respiratory, thoracic and mediastinal disorders) | 1
dry mouth (Gastrointestinal disorders) | 60
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Dsyphagia (Gastrointestinal disorders) | 1
DVT (Vascular disorders) | 1
dypsnea (Respiratory, thoracic and mediastinal disorders) | 2
Dysesthesia (Nervous system disorders) | 1
dysgeusia (Nervous system disorders) | 65
Dyspepsia (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 63
dysphonia (General disorders) | 5
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
dysuria (Renal and urinary disorders) | 4
ear ache (Ear and labyrinth disorders) | 1
ear congestion (Ear and labyrinth disorders) | 2
Ear disorder - other (Ear and labyrinth disorders) | 1
Ear infection (Ear and labyrinth disorders) | 2
ear pain (Ear and labyrinth disorders) | 17
easy bruising (Vascular disorders) | 2
Edema (General disorders) | 13
Edema limbs (General disorders) | 1
elbow pain (General disorders) | 1
elevated ANC (Investigations) | 1
elevated bilirubin (Investigations) | 2
elevated CO2 (Investigations) | 1
elevated creatinine (Investigations) | 10
Elevated prothrombin (Investigations) | 1
elevated WBC (Investigations) | 1
emesis (Hepatobiliary disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
erythema (Skin and subcutaneous tissue disorders) | 21
esophagitis (Gastrointestinal disorders) | 1
eye disorder- other (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Eye redness (Eye disorders) | 1 (1)
Facial edema (General disorders) | 1 (2)
Facial rash (Skin and subcutaneous tissue disorders) | 4 (4)
Facial swelling (General disorders) | 2 (2)
Factor V (Blood and lymphatic system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 11 (13)
Fatigue (General disorders) | 58 (103)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 12 (17)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Focal weakness (Nervous system disorders) | 2 (2)
Foot pain (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 3 (3)
G tube dysfunction (Gastrointestinal disorders) | 3 (3)
G tube placement (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - other, melena (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 2 (2)
Generalized weakness (General disorders) | 17 (22)
GERD (Gastrointestinal disorders) | 2 (2)
Gingival ulceration (Gastrointestinal disorders) | 1 (1)
Hair loss (Skin and subcutaneous tissue disorders) | 8 (9)
Hallucinations (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 18 (27)
Hearing impaired (Ear and labyrinth disorders) | 2 (2)
Hearing loss (Ear and labyrinth disorders) | 13 (14)
Heartburn (Gastrointestinal disorders) | 2 (2)
Heat intolerance (General disorders) | 1 (1)
Hematochezia (rectal bleeding) (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hernia (Injury, poisoning and procedural complications) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
High cholesterol (Investigations) | 3 (3)
Hip pain (General disorders) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 21 (25)
Hot flashes (Vascular disorders) | 4 (5)
Hypochloride (Investigations) | 23 (52)
Hypercalcemia (Metabolism and nutrition disorders) | 8 (10)
Hyperchloride (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 22 (43)
Hyperkalemia (Metabolism and nutrition disorders) | 12 (18)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 3 (5)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 7 (7)
Hypersalivation (Gastrointestinal disorders) | 2 (3)
Hypertension (Vascular disorders) | 42 (88)
Hyperthyroid (Endocrine disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 (27)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (22)
Hypochloremia (Investigations) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 17 (32)
Hypomagnesemia (Metabolism and nutrition disorders) | 15 (24)
Hyponatremia (Metabolism and nutrition disorders) | 26 (54)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4)
Hypophosphorous (Investigations) | 2 (4)
Hypotension (Vascular disorders) | 12 (13)
Hypothyroidism (Endocrine disorders) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 7 (7)
Infections and infestations - other, COVID-19 (Infections and infestations) | 1 (1)
Inflammation (General disorders) | 1 (1)
Influenza (flu-like symptoms) (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Injury, other, (mild fall injury) (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 29 (32)
Itching (General disorders) | 3 (3)
Jaw Pain (General disorders) | 6 (7)
Jaw Spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 11 (12)
Knee pain (Musculoskeletal and connective tissue disorders) | 2 (2)
L Elbow Pain (Metabolism and nutrition disorders) | 1 (1)
L knee pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal Edema (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Laryngitis (Infections and infestations) | 1 (1)
LE edema (General disorders) | 4 (4)
Leukocytosis (Investigations) | 5 (6)
Leukopenia (Investigations) | 1 (2)
Leukoplakia (General disorders) | 2 (2)
Localized edema (General disorders) | 23 (30)
Loss of smell (General disorders) | 8 (9)
Low total protein (General disorders) | 1 (1)
Lower extremity pain (General disorders) | 1 (1)
Lumbar stenosis (Nervous system disorders) | 1 (1)
Lump on abdomen (General disorders) | 1 (1)
Lung infection (Injury, poisoning and procedural complications) | 5 (5)
Lymphadenopathy (General disorders) | 2 (2)
Lymphadema (General disorders) | 30 (32)
Lymphocyte count decreased (Investigations) | 51 (194)
Macular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Mediastinal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Memory loss (Nervous system disorders) | 1 (1)
Mental confusion (Psychiatric disorders) | 1 (1)
Middle-ear infection (Ear and labyrinth disorders) | 1 (1)
Migraines (General disorders) | 1 (1)
Mild odynophagia (Gastrointestinal disorders) | 1 (1)
Mouth pain (Gastrointestinal disorders) | 1 (1)
Mouth sores (Gastrointestinal disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis (Gastrointestinal disorders) | 26 (47)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder - other (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgias (Musculoskeletal and connective tissue disorders) | 11 (13)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 22 (25)
Nausea (Gastrointestinal disorders) | 50 (97)
Neck edema (General disorders) | 6 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 39 (58)
Neoplasms benign - other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Nervous system disorder - other (Nervous system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 16 (30)
Neutrophil count increased (Investigations) | 7 (13)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4)
Nocturia (Renal and urinary disorders) | 7 (7)
Nocturnal "sweats" (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Nose bleeds (General disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 65 (148)
Oral dysesthesia (Nervous system disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral lesions (Gastrointestinal disorders) | 1 (1)
Oral mucositis (Gastrointestinal disorders) | 43 (88)
Oral pain (Gastrointestinal disorders) | 56 (124)
Oral thrush (Infections and infestations) | 2 (2)
Oropharyngeal edema (General disorders) | 1 (1)
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Otalgia (Ear and labyrinth disorders) | 1 (2)
Otic pain (L ear) (Ear and labyrinth disorders) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Pain (General disorders) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2)
Pallor (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (2)
Parathesia (Nervous system disorders) | 5 (6)
Peripheral neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (2)
Platelet count decreased (Investigations) | 31 (54)
Platelet count increased (Investigations) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Polydipsia (General disorders) | 6 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 31 (42)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Pulmonary embolism (Vascular disorders) | 1 (1)
R Otalgia (Ear and labyrinth disorders) | 1 (1)
Radiation dermatitis (Skin and subcutaneous tissue disorders) | 64 (114)
Radiation ulceration (Injury, poisoning and procedural complications) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 14 (19)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
rectal bleeding (Gastrointestinal disorders) | 1 (1)
rectal fissue (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Red eyes (Eye disorders) | 1 (1)
Reflux (Gastrointestinal disorders) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 1 (1)
Respiratory disorder- other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhonchus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rib pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right arm pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right chin pain (General disorders) | 1 (1)
Right ear pain (Ear and labyrinth disorders) | 1 (1)
Right eye pain (Eye disorders) | 1 (1)
Right inguinal hernia (Injury, poisoning and procedural complications) | 1 (1)
Right jaw pain (General disorders) | 1 (1)
Saliva pooling (Gastrointestinal disorders) | 1 (1)
Salivary duct inflammation (Gastrointestinal disorders) | 4 (6)
Salivary inflammation (Gastrointestinal disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Seasonal allergies (General disorders) | 8 (8)
Sensory change (General disorders) | 6 (7)
Sexual dysfunction (Reproductive system and breast disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Sinus pressure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder- other (Skin and subcutaneous tissue disorders) | 3 (3)
Skin erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5 (6)
Skin infection (Infections and infestations) | 2 (2)
Skin pigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Snoring (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 52 (127)
Speech change (General disorders) | 2 (2)
Stoma site infection (Infections and infestations) | 1 (1)
Stomal pain (General disorders) | 4 (6)
Stridor (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Surgical Procedure - other (Surgical and medical procedures) | 10 (10)
Syncope (Nervous system disorders) | 3 (3)
Syncopal (Nervous system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 8 (10)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 2 (2)
Thick saliva (Gastrointestinal disorders) | 7 (7)
Thick secretions (General disorders) | 49 (83)
Throat pain (Respiratory, thoracic and mediastinal disorders) | 12 (15)
Thrush (Infections and infestations) | 37 (50)
Tinnitus (Ear and labyrinth disorders) | 20 (28)
Toothache (Gastrointestinal disorders) | 2 (2)
Total bilirubin elevated (Investigations) | 1 (1)
Total protein decreased (Investigations) | 1 (1)
Tracheitis (Infections and infestations) | 1 (4)
Tremors (Nervous system disorders) | 3 (3)
Trismus (Musculoskeletal and connective tissue disorders) | 7 (7)
TSH elevated (Investigations) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ulceration (Injury, poisoning and procedural complications) | 5 (6)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 12 (12)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (6)
Urinary urgency (Renal and urinary disorders) | 7 (7)
Urine output decreased (Renal and urinary disorders) | 1 (1)
Velopharyngeal insufficiency (VPI) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 14 (15)
Vomiting (Gastrointestinal disorders) | 26 (46)
Weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Weight gain (Investigations) | 6 (6)
Weight loss (Investigations) | 61 (119)
wheezing (Respiratory, thoracic and mediastinal disorders) | 8 (8)
White blood cell count increased (Investigations) | 8 (12)
White blood cell count decreased (Investigations) | 36 (93)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Xerostomia (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT03067610/Prot_SAP_000.pdf